CLINICAL TRIAL: NCT01216332
Title: Randomized, Double Blind, Comparison of Standard Dose Trivalent Inactivated Influenza Vaccine Versus High Dose Trivalent Inactivated Influenza Vaccine in Pediatric Patients With Acute Lymphoblastic Leukemia
Brief Title: Standard Versus High-Dose Trivalent Inactivated Flu Vaccine in Pediatric Acute Lymphoblastic Leukemia Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Natasha Halasa, Assistant Professor, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VICC PED 1067
Record Dates: First submitted 2010-10-05; First posted 2010-10-07 (Estimated); Results first posted 2019-05-03 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-04

CONDITIONS: Pediatric Patients With Acute Lymphoblastic Leukemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High-Dose trivalent inactivated influenza vaccine (Experimental): 0.5 mL of high-dose trivalent inactivated influenza vaccine, either one dose or 2 based on whether the patient has previously received standard dose trivalent inactivated influenza vaccine.
  Interventions: Drug: High-dose trivalent inactivated influenza vaccine
- Standard dose trivalent inactivated influenza vaccine (Active Comparator): 0.5 mL standard dose trivalent inactivated influenza vaccine, either one dose or 2 based on whether the patient has previously received standard dose trivalent inactivated influenza vaccine
  Interventions: Drug: Standard dose trivalent inactivated influenza vaccine

INTERVENTIONS:
Drug: High-dose trivalent inactivated influenza vaccine — 0.5 mL of high-dose trivalent inactivated influenza vaccine, either one dose or 2 based on whether the patient has previously received standard dose trivalent inactivated influenza vaccine.
  Arms: High-Dose trivalent inactivated influenza vaccine
Drug: Standard dose trivalent inactivated influenza vaccine — 0.5 mL standard dose trivalent inactivated influenza vaccine
  Arms: Standard dose trivalent inactivated influenza vaccine

SUMMARY:
This is a phase I safety and immunogenicity trial comparing high-dose (HD)trivalent inactivated influenza vaccine (TIV) to standard dose (SD) TIV in pediatric patients with Acute Lymphoblastic Leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients with standard or high risk Acute Lymphoblastic Leukemia.
* Must be in 1st complete remission.
* Must be 4 weeks into maintenance therapy.
* 17 years of age, inclusive.
* Available for duration of study.

Exclusion Criteria:

* History of hypersensitivity to previous influenza vaccination or hypersensitivity to eggs/egg protein.
* History of Guillain-Barre syndrome.
* Evidence of relapsed disease.
* Have any condition that would, in the opinion of the site investigator, place them at an unacceptable risk of injury or render them unable to meet the requirements of the protocol.
* Have any condition that the investigator believes may interfere with successful completion of the study.
* History of receiving 2010 - 2011 influenza vaccine.
* Pregnant female.
* History of proven influenza disease after September 1, 2010.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2010-10; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natasha Halasa, M.D., Principal Investigator — Vanderbilt Universtiy Medical Center
Locations (1):
- Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Four subjects (from the high dose group) were excluded from the data analysis , because they were given the second dose of TIV outside the study window period. These four subjects were included in the adverse event reporting.
Period: Overall Study
Arm/Group | High-Dose Trivalent Inactivated Influenza Vaccine | Standard Dose Trivalent Inactivated Influenza Vaccine
Started | 34 | 16
Completed | 30 | 16
Not Completed | 4 | 0
Not completed — Withdrawal by Subject | 4 | 0

BASELINE CHARACTERISTICS:
Population: Four subjects were excluded from the data analysis (from the high dose group), because they were given the second dose of TIV outside the study window period
Groups:
- Total: Total of all reporting groups
Arm/Group | High-Dose Trivalent Inactivated Influenza Vaccine | Standard Dose Trivalent Inactivated Influenza Vaccine | Total
Number analyzed (Participants) | 30 | 16 | 46
Age, Customized [Count of Participants; unit: Participants]
  <=18 years | 30 | 16 | 46
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 12 | 5 | 17
  Male | 18 | 11 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 28 | 12 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 27 | 12 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 16 | 46

OUTCOME MEASURES:

1. Primary Outcome: Local Reactions After Each Vaccination
Description: Number of participants with local reactions after each vaccination
Time Frame: From baseline to 7 days after each vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | High-Dose Trivalent Inactivated Influenza Vaccine | Standard Dose Trivalent Inactivated Influenza Vaccine
Number analyzed (Participants) | 30 | 16
Participants
  Pain | 12 | 7
  Tenderness | 14 | 9
  Intense Swelling | 3 | 3
  Redness | 4 | 2

2. Primary Outcome: Systemic Reaction
Description: Number of participants with systemic reactions after each vaccination
Time Frame: From baseline to 7 days after each vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | High-Dose Trivalent Inactivated Influenza Vaccine | Standard Dose Trivalent Inactivated Influenza Vaccine
Number analyzed (Participants) | 30 | 16
Participants
  Fatigue | 14 | 14
  Decrease in Activity | 13 | 7
  Fever | 4 | 3
  Headache | 6 | 9
  Nausea | 7 | 6
  Body aches | 6 | 3
  Vomiting | 2 | 7

3. Secondary Outcome: Immunogenicity: Number of Participants With a Post-titer Greater Than or Equal to a Fourfold Titer Rise
Description: Greater than or equal to a Fourfold titer rise three strains (A/California/7/09/H1N1, A/Perth/16/2009/ H3N2, B/Brisbane/60/2008)
Time Frame: About 6 months after last dose of vaccine.
Population: Participants that receive only 1 dose of vaccine. In addition, two subjects were excluded due to lack of complete immunogenicity data
Measure: Count of Participants; unit: Participants
Arm/Group | High-Dose Trivalent Inactivated Influenza Vaccine | Standard Dose Trivalent Inactivated Influenza Vaccine
Number analyzed (Participants) | 24 | 13
Participants
  A/California/7/09 H1N1 | 6 | 6
  A/Perth/16/2009 H3N2 | 8 | 5
  B/Brisbane/60/2008 | 2 | 0

4. Secondary Outcome: Immunogenicity:Number of Participants With a Pre-titer ≥1:40
Description: Pre-titer ≥1:40 for three strains (A/California/7/09/H1N1, A/Perth/16/2009/ H3N2, B/Brisbane/60/2008)
Time Frame: About 6 months after last dose of vaccine.
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | High-Dose Trivalent Inactivated Influenza Vaccine | Standard Dose Trivalent Inactivated Influenza Vaccine
Number analyzed (Participants) | 24 | 13
Participants
  A/California/7/09 H1N1 | 17 | 9
  A/Perth/16/2009 H3N2 | 9 | 7
  B/Brisbane/60/2008 | 21 | 11

5. Secondary Outcome: Immunogenicity: Number of Participants With a Post-titer ≥1:40
Description: Post-titer ≥1:40 for three strains (A/California/7/09/H1N1, A/Perth/16/2009/ H3N2, B/Brisbane/60/2008)
Time Frame: About 6 months after last dose of vaccine.
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | High-Dose Trivalent Inactivated Influenza Vaccine | Standard Dose Trivalent Inactivated Influenza Vaccine
Number analyzed (Participants) | 24 | 13
Participants
  A/California/7/09 H1N1 | 20 | 11
  A/Perth/16/2009 H3N2 | 13 | 8
  B/Brisbane/60/2008 | 19 | 9

6. Secondary Outcome: Immunogenicity: The Geometric Mean Titers Pre-vaccine in Study Participants
Description: Geometric mean titers pre-vaccine (A/California/7/09/H1N1, A/Perth/16/2009/ H3N2, B/Brisbane/60/2008)
Time Frame: baseline
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | High-Dose Trivalent Inactivated Influenza Vaccine | Standard Dose Trivalent Inactivated Influenza Vaccine
Number analyzed (Participants) | 24 | 13
Titers
  A/California/7/09 H1N1 | 46.2 [27.4 to 75.7] | 87.4 [37.9 to 209.1]
  A/Perth/16/2009 H3N2 | 28.3 [18.7 to 43.3] | 28.8 [18.1 to 46.5]
  B/Brisbane/60/2008 | 66.5 [51.8 to 82.2] | 56.1 [43.9 to 69.4]

7. Secondary Outcome: Immunogenicity: Geometric Mean Titers Post-vaccine in Study Participants
Description: Geometric mean titers post-vaccine (A/California/7/09/H1N1, A/Perth/16/2009/ H3N2, B/Brisbane/60/2008)
Time Frame: About 6 months after last dose of vaccine.
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | High-Dose Trivalent Inactivated Influenza Vaccine | Standard Dose Trivalent Inactivated Influenza Vaccine
Number analyzed (Participants) | 24 | 13
Titers
  A/California/7/09 H1N1 | 97.9 [61.1 to 166.3] | 322.9 [141.3 to 792.1]
  A/Perth/16/2009 H3N2 | 62.9 [34.6 to 122.2] | 76.5 [36 to 176.5]
  B/Brisbane/60/2008 | 74.4 [49.9 to 111.6] | 50.6 [35.3 to 67.3]

ADVERSE EVENTS:
Time Frame: AEs were collected for 28 days after last vaccination, and SAEs were collected through 180 days after their final vaccination via phone call and medical chart review.
Arm/Group | High-Dose Trivalent Inactivated Influenza Vaccine | Standard Dose Trivalent Inactivated Influenza Vaccine
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/16
Serious Adverse Events (participants affected / at risk) | 9/34 | 6/16
Other Adverse Events (participants affected / at risk) | 21/34 | 14/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High-Dose Trivalent Inactivated Influenza Vaccine (N=34) | Standard Dose Trivalent Inactivated Influenza Vaccine (N=16)
Acute Otitis Media (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Influenza B (Infections and infestations) | 0 (0) | 2 (2)
Fever (General disorders) | 4 (5) | 0 (0)
Coronavirus (Infections and infestations) | 1 (2) | 0 (0)
Viral Illness (Infections and infestations) | 2 (2) | 2 (2)
New Onset Seizures (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High-Dose Trivalent Inactivated Influenza Vaccine (N=34) | Standard Dose Trivalent Inactivated Influenza Vaccine (N=16)
Redness at injection site (General disorders) | 4 | 2
Pain at Injection Site (General disorders) | 12 | 3
Tenderness (General disorders) | 14 | 9
Intense Swelling (General disorders) | 3 | 3
Fatigue (General disorders) | 14 | 14
Decrease in Activity (General disorders) | 13 | 7
Fever (General disorders) | 4 | 3
Headache (General disorders) | 6 | 9
Nausea (General disorders) | 7 | 6
Body Aches (General disorders) | 6 | 3
Vomiting (General disorders) | 2 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No